CLINICAL TRIAL: NCT05674266
Title: New Treatment Perspectives in Adolescents With Anorexia Nervosa: the Efficacy of Non-invasive Brain-directed Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 763_OPBG_2014_BIS
Record Dates: First submitted 2022-12-06; First posted 2023-01-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Anorexia in Adolescence
Keywords: tDCS; EEG; TMS; cortisol; eating disorder; neuromodulation
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AN Active tDCS (Experimental): Treatment "as usual" plus experimental treatment
  Interventions: Device: AN Active tDCS
- AN Sham tDCS (Sham Comparator): Treatment "as usual" plus placebo treatment
  Interventions: Device: AN Sham tDCS

INTERVENTIONS:
Device: AN Active tDCS — The tDCS active stimulations will be directed to PFC regions for six weeks delivered for three times a week.
  tDCS will be delivered by a battery driven, constant current stimulator through a pair of saline-soaked sponge electrodes kept firm by elastic bands.
  The anode will be placed on the left PFC, F3 position according to the 10-20 international EEG system for electrode placement, while the cathode will be placed on the right PFC, F4 position according to the 10-20 international EEG system for electrode placement.
  Stimulation intensity will be set at 1 milliampere (mA), the duration of stimulation will be 20 min.
  Other Names: Brain Stim
  Arms: AN Active tDCS
Device: AN Sham tDCS — The same electrode placement will be used as in the stimulation conditions (left anodal/right cathodal), but the current will be applied for 30 s and will be ramped down without the participants awareness, and will be held three times a week for six weeks.
  Other Names: Brain Stim Sham
  Arms: AN Sham tDCS

SUMMARY:
The present randomized, double blind, placebo-controlled trial aims at evaluating the efficacy of a tDCS treatment in improving the clinical outcome of adolescents with AN and investigate brain mechanisms acting in AN.

DETAILED DESCRIPTION:
The investigators hypothesized that excitatory tDCS over the left PFC and inhibitory tDCS over the right PFC (anode left/cathode right) may aid in altering/resetting inter-hemispheric balance in children and adolescents with AN, reducing their control over eating behaviors and improving the AN psychopathology. Furthermore, the investigators will employ TMS-EEG to directly explore the DLPFC activity of children and adolescent with AN, with specific attention to the differences between hemispheres. Moreover, paired pulse TMS and repetitive TMS protocols will be used to investigate the functional mechanisms within the prefrontal cortex of youth patients with AN. Then, the investigators will assess if potential changes of specific biomarkers, such as those related to the endogenous stress response system functioning, will occur after tDCS treatment and will correlate with clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of AN according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition - DSM-5 (American Psychiatric Association & American Psychiatric Association, 2013);
* condition of under-weight (BMI <18.5 kg/m2);
* intelligence quotient higher or equal to 85 (IQ ≥ 85);
* ability to give informed consent under parents' surveillance and guidance

Exclusion Criteria:

* a personal history of neurological/medical/genetic diseases;
* a personal history of epilepsy;
* suicide risk;
* receiving CNS-active drug, other counseling or psychological therapies during the treatment.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
The primary end-point of the study is the variance on eating psychopathology at T1, assessed as changes in Eating Disorder Risk score (EDRC) of the Eating Disorder Inventory (EDI-3). Significant changes in Ineffectiveness (IC) of the EDI-3. | 6 weeks
  EDI-3 comprises 91-item that give a measure of the basic characteristics of the ED through six composite scores [Eating Disorder Risk (EDRC) (range 0-100), Ineffectiveness (IC) (range 0-48), Interpersonal Problems (IPC) (range 0-52), Affective Problems (APC) (range 0-62), Overcontrol (OC) (range 0-52), and General Psychological Maladjustment (GPMC) (range 0-252)]. Higher scores indicates more severe problems.

SECONDARY OUTCOMES:
Significant changes in Ineffectiveness (IC) of the EDI-3. | 12 months follow up
  Evaluation of the change in Ineffectiveness, with maximum possible score of 48, where higher scores indicate higher Ineffectiveness.
Significant changes in Interpersonal Problems (IPC) of the EDI-3. | 12 months follow up
  Evaluation of the change in Interpersonal Problems, with maximum possible score of 52, where higher scores indicate higher Interpersonal Problems.
Significant changes in Affective Problems (APC) of the EDI-3. | 12 months follow up
  Evaluation of the change in Affective Problems, with maximum possible score of 62, where higher scores indicate higher Affective Problems.
Significant changes in Overcontrol (OC) of the EDI-3. | 12 months follow up
  Evaluation of the change in Overcontrol, with maximum possible score of 52, where higher scores indicate higher Overcontrol.
Significant changes in General Psychological Maladjustment (GPMC) of the EDI-3. | 12 months follow up
  Evaluation of the change in General Psychological Maladjustment, with maximum possible score of 252, where higher scores indicate higher General Psychological Maladjustment.
Significant changes in the total scores of AN symptomatology measures as Eating Attitudes Test (EAT-26) | 12 months follow up
  The EAT-26 proposes a cut-off score of 20. Scores of 20 or higher were considered clinically significant.
Significant changes in the total scores of AN symptomatology measures as Body Uneasiness Test (BUT). | 12 months follow up
  The BUT proposes a cut-off score of 1,2. Scores of 1,2 or higher were considered clinically significant.
Significant changes in the total scores of other psychopathological measures as Child Behavior Checklist (CBCL 6-18). | 12 months follow up
  The CBCL 6-18 generates a T-score for each subscale. According to normative data, a T-score above 64 was considered to be significant for the 3 broadband scales, whereas for the syndrome scales, the cut-off for clinical significance was 70.
Significant changes in the total scores of other psychopathological measures as Children's Depression Inventory (CDI). | 12 months follow up
  Raw scores were converted to T-scores. According to normative data, a T-score above 64 was considered clinical significance.
Significant changes in the total scores of other psychopathological measures as Multidimensional Anxiety Scale for Children (MASC). | 12 months follow up
  Raw scores were converted to T-scores. According to normative data, a T-score above 64 was considered clinical significance.
Significant changes in the physiological measures specifically the BMI index | 12 months follow up
Number of participants with abnormal laboratory blood test results. | 12 months follow up
Significant changes in the endogenous stress response, measured with Cortisol Awakening Response (CAR). | 12 months follow up
Significant changes in intra-cortical inhibitory/excitatory motor circuits using paired pulse TMS, measured as short intracortical inhibition and facilitation. | 6 weeks
  the ratio between MEPs amplitude conditioning stimulus and MEPs amplitude test stimulus alone for each ISI.
Significant changes in sensory-motor integration using paired pulse TMS, measured as SICI/ICF: the ratio between MEPs amplitude (mV) conditioning stimulus (electrical stimulation) and MEP amplitude test stimulus alone for each ISI. | 6 weeks
Significant changes in cortical oscillatory patterns (synchronization and desynchronization) in theta, alpha and beta frequencies (Hz) over motor and premotor cortex, using TMS-EEG co-registration. | 6 weeks
Significant changes in cortical connectivity using TMS-EEG co-registration combined to report the analysis of the waveform, latency and cortical distribution of TMS-evoked potentials (TEPs) in micronV. | 6 weeks
Significant changes in cortical reactivity in terms of TMS-evoked potentials (TEPs) amplitude for time domain (micronV) and frequency bands for spatial domain (Hz), using TMS-EEG co-registration. | 6 weeks
Significant changes in Cortical Plasticity evoked by repetitive TMS in terms of different MEP amplitude (mV) recorded at different time-points after repetitive TMS perturbations. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Floriana Costanzo, Principal Investigator — Bambino Gesù Hospital and Research Institute; Stefano Vicari, Study Chair — Bambino Gesù Hospital and Research Institute
Locations (1):
- Bambino Gesù Hospital and Research Institute, Rome, Italy

REFERENCES:
- [Background] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Result] Costanzo F, Menghini D, Maritato A, Castiglioni MC, Mereu A, Varuzza C, Zanna V, Vicari S. New Treatment Perspectives in Adolescents With Anorexia Nervosa: The Efficacy of Non-invasive Brain-Directed Treatment. Front Behav Neurosci. 2018 Jul 20;12:133. doi: 10.3389/fnbeh.2018.00133. eCollection 2018. PMID 30083095
- [Derived] Ursumando L, Ponzo V, Monteleone AM, Menghini D, Fuca E, Lazzaro G, Esposito R, Picazio S, Koch G, Zanna V, Vicari S, Costanzo F. The efficacy of non-invasive brain stimulation in the treatment of children and adolescents with Anorexia Nervosa: study protocol of a randomized, double blind, placebo-controlled trial. J Eat Disord. 2023 Aug 2;11(1):127. doi: 10.1186/s40337-023-00852-6. PMID 37533058